CLINICAL TRIAL: NCT04232007
Title: Closed-loop Control of Vasopressor Administration in High-Risk Patients Undergoing Cardiac Surgery: A Case Series
Brief Title: Closed-loop Control of Vasopressor Administration in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Collaborators: University of California, Los Angeles (Other); University of California, Irvine (Other)
Responsible Party: Principal Investigator, Alexandre Joosten, MD PhD, Principal Investigator, Erasme University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P2018(276)
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Hemodynamic MAP Stability

STUDY DESIGN:
Intervention Model Description: Closed-loop system to titrate vasopressor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Closed-loop (Experimental): Closed-loop system to titrate vasopressor during surgery
  Interventions: Device: closed-loop system for vasopressor administration

INTERVENTIONS:
Device: closed-loop system for vasopressor administration — closed-loop system for vasopressor administration

SUMMARY:
Intraoperative hypotension and blood pressure variability are associated with postoperative complications in surgical patients.

The investigators have developed a closed-loop vasopressor (CLV) controller that titrates norepinephrine to correct hypotension.

After having tested the system in a small cohort series of patients undergoing major surgeries, the investigators aimed to test the feasibility of the CLV controller in three high risk patients undergoing cardiac surgery

DETAILED DESCRIPTION:
The investigators have recently developed an automated closed-loop vasopressor (CLV) controller to better titrate vasopressor (e.g:norepinephrine) to maintain MAP within a narrow range (±5mmHg of the chosen target).

The investigators published engineering, animal studies and recently described the feasibility of titration of norepinephrine in 20 patients undergoing major noncardiac procedures. This initial cohort human study showed the controller was able to keep patients within ± 5 mmHg of a target pressure for more than 90% of management time. Cardiac surgery represents unique challenges in MAP management as the manipulation of the heart itself, the use of cardiopulmonary bypass (CPB) and cardioplegia, and the pre-existing cardiac disease all increase the difficulty in maintaining a steady MAP throughout the surgical period.

In this case series the investigators describe three cardiac surgical procedures managed with the CLV system (one coronary artery bypass graft (CABG) procedure done under CPB; one robotic minimally invasive direct coronary artery bypass (MIDCAB) procedure (through a mini-thoracotomy), and one off-pump CABG) in order to assess its feasibility, efficiency and behavior in three high-risk patients before starting a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult high risk patients undergoing cardiac surgery (robotic, off-pump and on pump cardiac surgery)

Exclusion Criteria:

* Atrial fibrillation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
percentage of time spent during surgery in hypotension | during surgery
  percentage of time spent during surgery in hypotension defined as a MAP below 65 mmHg.

SECONDARY OUTCOMES:
time in target during surgery | during surgery
  time with a MAP within 5 mmHg of the chosen target
Percentage of active treatment time spent in a hypertensive state | during surgery
  Percentage of active treatment time spent in a hypertensive state, defined as a MAP >5mmHg above the chosen target MAP with an active norepinephrine infusion
Amount of vasopressor used | during surgery
  Amount of vasopressor administered to the patient

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Joosten, Principal Investigator — ERASME
Locations (1):
- Erasme, Brussels, Anderlecht, Belgium

IPD SHARING:
Plan to Share IPD: No